CLINICAL TRIAL: NCT02067858
Title: An Outcome Analysis for Stereotactic Body Radiation Therapy (SBRT) Treatment of Non-Small Lung Cancer Patients Using 4D PET/CT With Real-Time Position Management (RPM™) System and a Concomitant Evaluation of the Impact and Performance Characteristics of the Immobilization System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: Steven Burton (Other)
Responsible Party: Sponsor-Investigator, Steven Burton, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10-003
Record Dates: First submitted 2014-02-14; First posted 2014-02-20 (Estimated); Results first posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-06

CONDITIONS: Non Small Cell Lung Cancer; 4D CT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic Radiosurgery (Other): 3 fractions x 20 Gy 4 fractions x 12 Gy
  Lesion dependent
  Interventions: Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery
  Other Names: SBRT; SRS; Trilogy; True Beam; Cyber Knife

SUMMARY:
The goals of this clinical research are to evaluate the outcomes and tumor response for early stage non-small lung cancer (NSCLC) patients undergoing Stereotactic Body Radiation Therapy (SBRT) using four dimensional (4D) Positron Emission Tomography (PET) and Computed Tomography (CT), Cone-Beam Computed Tomography (CBCT), Real-Time Position Management (RPM™) and body immobilization system (see figure 1). Specifically, the effect of image-guided SBRT treatment on clinical tumor response rate, local control and progression-free survival will be studied. This study will examine target volumes and relevant margins determined by an assessment using 4D PET and repeated 4D CT. These data will allow us to evaluate and determine the impact of the body immobilization system on the planning target volume (PTV) margins, patient's breathing pattern, target motion, and inter-treatment targets shifts.

ELIGIBILITY:
The patient must be over the age of 18 years. Histologic confirmation of primary NSCLC of the lung tumor must be complete prior to SBRT treatment.

The following stages of NSCLC patients would be eligible for the study:

Stage I:

T1 N0 M0 T2 N0 M0 (Size ≤ 5 cm)

Stage II:

T3 N0 M0 (Chest wall invasion only, Size ≤ 5 cm)

Staging Tumor size and characteristics: they will be determined by PET-CT scan

Nodal disease:

Patients with chest CT scan demonstrating hilar or mediastinal nodes <1cm and/or PET negative would be considered N0 disease.

Patients who have hilar or mediastinal nodes > 1 cm and PET scan negative may be considered N0 disease.

If PET scan demonstrates suspicious uptake or abnormal uptake, these patients would be eligible, if a directed biopsy (by mediastinoscopy, Chamberlein procedure or other modalities such as trans-bronchial biopsy, CT guided biopsy) is negative.

Metastases:

Evaluated by PET-CT scanning and biopsy as indicated

The patient must have an ECOG/Zubrod performance status of 0, 1, or 2. In order to be considered medically-inoperable, the patient must meet at least one major criterion or meet a minimum of 2 minor criteria as described below.

MAJOR CRITERIA:

FEV1 < 50% or predicted postoperative FEV1 < 40% DLCO < 50% or predicted postoperative DLCO < 40% Exercise induced maximal exercise oxygen consumption (MVO2)<15 ml/kg/min Thoracic surgery consultation should be obtained from a Board Certified Thoracic surgeon who in collaboration with a radiation oncologist should determine if the patient is medically operable This criterion would be mandatory

MINOR CRITERIA:

Age > 80 Pulmonary hypertension (defined as a pulmonary artery systolic pressure greater than 40mm Hg) Oxygen requirement (using the Medicare criteria for home oxygen requirements [i.e., room air oxygen saturation of 88% or less]) Congestive heart failure (any three of the following must be documented: dyspnea, peripheral edema, chest x-ray with interstitial edema or cardiomegaly, rales, or congestion) Poor left ventricular function (defined as an ejection fraction of 40% or less) Severe cerebral (with CVA or recent TIA) or severe peripheral vascular disease Diabetes Mellitus with severe organ damage such as End-Stage Renal Disease (ESRD), Blindness, Vascular disease.

CBC, Diff and platelets, Comprehensive metabolic panel within 28 days of registration meeting the following criteria

leukocytes >3,000/mcL absolute neutrophil count >1,500/mcL hemoglobin >9 g/dL (hemoglobin may be supported by transfusion or erythropoietin or other approved hematopoietic growth factors) platelets >100,000/mcL total bilirubin <1.5x institutional upper limit of normal creatinine within normal institutional limits OR creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.

Females of child-bearing age must be using a reliable form of birth control. The patient must provide a signed and dated written informed consent PRIOR to registration and prior to undergoing any study-related procedures.

The patient must provide written authorization to allow for the use and disclosure of their protected Health information.

Conditions for Patient Ineligibility The patient's weight exceeds the tolerances of the institution's imaging and treatment platform/couch.

The patient has received thoracic radiation therapy in the same region as the current SBRT planned treatment area. The patient has completed chemotherapy within 30 days of treatment. T2: Tumor size > 5 cm, T3 tumors (except T3 by virtue of chest wall invasion and ≤ 5cm), T4 tumors. Presence of N1, N2 or N3 disease per previously described criteria would also be excluded.

Pancoast tumors would be excluded. Current distant metastatic disease (M1) (preferably biopsy proven). The patient is a female with child-bearing potential who refuses to obtain a serum pregnancy test prior to the initiation of treatment.

The patient is pregnant or a female who is nursing an infant. The patient is planning on undergoing systemic therapy within 2 weeks after the last fraction of radiation The patient has an active systemic or pulmonary infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dwight E Heron, MD, Study Chair — University of Pittsburgh
Locations (1):
- UPMC Shadyside Radiation Oncology Department, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Stereotactic Radiosurgery: 3 fractions x 20 Gy 4 fractions x 12 Gy
  Lesion dependent
  Stereotactic Radiosurgery
Period: Overall Study
Arm/Group | Stereotactic Radiosurgery
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Assess Clinical Response Rate and Local Control Following SBRT Treatment of Patients With Early Stage NSCLC
Description: The Number of Patients that completed SBRT
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 6
Participants | 4

2. Secondary Outcome: Assess Progression-free Survival
Description: Number of patients with Progression Free Survival at 2 Years
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 3
Participants | 3

3. Other Pre Specified Outcome: Correlation of Imaging Response With Serum Protein and Peptide Profiles
Description: Research blood draws looking at imaging repsonse before and after radiation in relationship to serum protein and peptide profiles
Time Frame: 2 years
Population: Blood draw samples were not drawn nor analyzed for this study
Arm/Group | Stereotactic Radiosurgery
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Stereotactic Radiosurgery
All-Cause Mortality (participants affected / at risk) | 5/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes